CLINICAL TRIAL: NCT06241820
Title: The Success of Lumbar Sympathetic Ganglion Block Using Lower Extremity Perfusion Index: A Prospective Observational Study
Brief Title: The Success of Lumbar Sympathetic Ganglion Block Using Lower Extremity Perfusion Index
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jeongsoo Kim (Other)
Responsible Party: Sponsor-Investigator, Jeongsoo Kim, Professor, Seoul National University Hospital
Organization: Seoul National University Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2308-014-1455
Record Dates: First submitted 2024-01-28; First posted 2024-02-05 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Chronic Pain; Complex Regional Pain Syndromes; Peripheral Neuropathy; Post Herpetic Neuralgia
MeSH Terms: conditions — Chronic Pain; Complex Regional Pain Syndromes; Peripheral Nervous System Diseases; Neuralgia, Postherpetic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lumbar Sympathetic Ganglion Block (LSGB) (Other): FS-guided LSGB at L3 level.
  Interventions: Procedure: Lumbar Sympathetic Ganglion Block

INTERVENTIONS:
Procedure: Lumbar Sympathetic Ganglion Block — A needle will be inserted at the L3 on the side experiencing pain, either right or left, under fluoroscopy guidance. Once the needle is positioned in front of the desired vertebral body, its location is confirmed using a contrast medium. If the position is well visualized in lateral and anteroposterior (AP) views, 7 mL of 0.5% ropivacaine will be injected.

SUMMARY:
The patient, who is experiencing chronic pain in the lower extremities persisting for more than three months, is scheduled to undergo lumbar sympathetic ganglion block. To evaluate the technical success of the sympathetic blockade, temperature and perfusion index (PI) will be measured at one-minute intervals over a 20-minute period before and after the procedure on the treated side and the opposite side foot. Additionally, other variables related to the procedure will be assessed before the procedure, after the procedure, before discharge, and during follow-up outpatient visits or phone surveys at 1 week and 1 month after the procedure.

DETAILED DESCRIPTION:
Patients aged 19 to 85 experiencing lower limb pain and scheduled to undergo lumbar sympathetic ganglion block at the Seoul National University Hospital Pain Center will be directly informed about the study, and their participation will be sought and registered. Continuous monitoring of electrocardiography, blood pressure, and pulse oximetry will be conducted before and after the procedure.

Upon admission to the pain center's operating room, the patient will assume a prone position. Thermometers will be attached to the soles of both feet, and perfusion index probes will be attached to the second toe on both sides. Using fluoroscopy guidance, a needle will be inserted at the painful side, either right or left, at the L3. After confirming the needle's position in front of the desired vertebral body using contrast medium in lateral and anteroposterior (AP) views, 7 mL of 0.5% ropivacaine will be injected. Baseline temperature and PI values will be recorded before drug administration, followed by recording every minute for 20 minutes after injection.

Other variables related to the procedure will be assessed before and after the procedure, before discharge, and through outpatient visits or phone surveys at one week after the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Lower extremity pain
* Pain for more than 3 months
* 19 - 85 years

Exclusion Criteria:

* If the patient refuses to undergo the procedure
* In the presence of vascular disorders in the lower extremities
* If the patient has previously undergone lumbar sympathetic ganglion removal or neurolysis
* When there are abnormalities in blood coagulation tests
* If there is a systemic infection or infection at the injection site
* In the presence of anatomical deformities at the injection site
* If the patient has allergies to the injected medication
* In other cases where the researcher deems the patient unsuitable for participation

Ages: 19 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-02-13 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
Difference of perfusion index (%) | before and 1 - 20 minutes after FS-guided lumbar sympathetic ganglion block
  Difference of perfusion index (%) between ipsilateral foot and contralateral foot

SECONDARY OUTCOMES:
Difference of temperature change (°C) | before and 1 - 20 minutes after FS-guided lumbar sympathetic ganglion block
  Difference of temperature change (°C) between ipsilateral foot and contralateral foot
Severity of pain | Time before block and 20 minutes, 1 week, 4 weeks after FS-guided lumbar sympathetic ganglion block ( The higher the score, the more severe the pain)
  11-point Numerical Rating Scale (NRS, 0-10)
Proportion of patients reaching ≥ 1.5°C rise | 20 minutes after FS-guided lumbar sympathetic ganglion block
  Proportion of patients reaching ≥ 1.5°C rise of temperature in the ipsilateral foot compared to the contralateral foot
Proportion of patients reaching ≥ 2.0°C rise | 20 minutes after FS-guided lumbar sympathetic ganglion block
  Proportion of patients reaching ≥ 2.0°C rise of temperature in the ipsilateral foot compared to initial temperature in the ipsilateral foot
Proportion of patients reaching ≥ 100% rise of perfusion index (%) | 1 - 20 minutes after FS-guided lumbar sympathetic ganglion block
  Proportion of patients reaching ≥ 100% rise of perfusion index (%) in the ipsilateral foot compared to the initial perfusion index (%) in the ipsilateral foot
Patient satisfaction | Time 20 minutes, 1 week, 4 weeks after FS-guided lumbar sympathetic ganglion block (The higher the score, the higher the satisfaction)
  Patient Global Impression of Change (1-5)

CONTACTS AND LOCATIONS:
Overall Officials: Jeongsoo Kim, MD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Day M. Sympathetic blocks: the evidence. Pain Pract. 2008 Mar-Apr;8(2):98-109. doi: 10.1111/j.1533-2500.2008.00177.x. PMID 18366465
- [Background] Joo EY, Kong YG, Lee J, Cho HS, Kim SH, Suh JH. Change in pulse transit time in the lower extremity after lumbar sympathetic ganglion block: an early indicator of successful block. J Int Med Res. 2017 Feb;45(1):203-210. doi: 10.1177/0300060516681398. Epub 2017 Jan 17. PMID 28222636
- [Background] Stevens RA, Stotz A, Kao TC, Powar M, Burgess S, Kleinman B. The relative increase in skin temperature after stellate ganglion block is predictive of a complete sympathectomy of the hand. Reg Anesth Pain Med. 1998 May-Jun;23(3):266-70. doi: 10.1016/s1098-7339(98)90053-0. PMID 9613538
- [Background] Kim ED, Yoo WJ, Lee YJ, Park HJ. Perfusion index as a tool to evaluate the efficacy of stellate ganglion block for complex regional pain syndrome. Clin Auton Res. 2019 Apr;29(2):257-259. doi: 10.1007/s10286-018-00585-6. Epub 2019 Jan 1. No abstract available. PMID 30600407
- [Background] Lee JY, Kim ED, Kim YN, Kim JS, Sim WS, Lee HJ, Park HJ, Park HJ. Correlation of Perfusion Index Change and Analgesic Efficacy in Transforaminal Block for Lumbosacral Radicular Pain. J Clin Med. 2019 Jan 7;8(1):51. doi: 10.3390/jcm8010051. PMID 30621004
- [Background] Abdelnasser A, Abdelhamid B, Elsonbaty A, Hasanin A, Rady A. Predicting successful supraclavicular brachial plexus block using pulse oximeter perfusion index. Br J Anaesth. 2017 Aug 1;119(2):276-280. doi: 10.1093/bja/aex166. PMID 28854539
- [Background] Yamazaki H, Nishiyama J, Suzuki T. Use of perfusion index from pulse oximetry to determine efficacy of stellate ganglion block. Local Reg Anesth. 2012;5:9-14. doi: 10.2147/LRA.S30257. Epub 2012 Mar 13. PMID 22915896
- [Background] Ginosar Y, Weiniger CF, Meroz Y, Kurz V, Bdolah-Abram T, Babchenko A, Nitzan M, Davidson EM. Pulse oximeter perfusion index as an early indicator of sympathectomy after epidural anesthesia. Acta Anaesthesiol Scand. 2009 Sep;53(8):1018-26. doi: 10.1111/j.1399-6576.2009.01968.x. Epub 2009 Apr 24. PMID 19397502
- [Background] Huang B, Sun K, Zhu Z, Zhou C, Wu Y, Zhang F, Yan M. Oximetry-derived perfusion index as an early indicator of CT-guided thoracic sympathetic blockade in palmar hyperhidrosis. Clin Radiol. 2013 Dec;68(12):1227-32. doi: 10.1016/j.crad.2013.07.003. Epub 2013 Aug 19. PMID 23969155
- [Background] Cheng J, Salmasi V, You J, Grille M, Yang D, Mascha EJ, Cheng OT, Zhao F, Rosenquist RW. Outcomes of Sympathetic Blocks in the Management of Complex Regional Pain Syndrome: A Retrospective Cohort Study. Anesthesiology. 2019 Oct;131(4):883-893. doi: 10.1097/ALN.0000000000002899. PMID 31365367
- [Background] Samen CDK, Sutton OM, Rice AE, Zaidi MA, Siddarthan IJ, Crimmel SD, Cohen SP. Correlation Between Temperature Rise After Sympathetic Block and Pain Relief in Patients with Complex Regional Pain Syndrome. Pain Med. 2022 Sep 30;23(10):1679-1689. doi: 10.1093/pm/pnac035. PMID 35234922
- [Background] Kim J, Yun M, Han AH, Pauzi MF, Jeong JH, Yoo Y, Moon JY. Thoracic sympathetic ganglion blocks: real-world outcomes in 207 chronic pain patients. Reg Anesth Pain Med. 2024 Jul 8;49(7):528-535. doi: 10.1136/rapm-2023-104624. PMID 37726196